CLINICAL TRIAL: NCT07239986
Title: An Open-label, Multicenter Phase 2 Clinical Study on the Efficacy and Safety of BB102 in Patients With Advanced or Unresectable FGF19-overexpressing Hepatocellular Carcinoma
Brief Title: A Phase 2 Study of BB102 in Patients With Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Broadenbio Ltd., Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BB102-HCC-II-01
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: hepatocellular carcinoma; FGFR4; BB102
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BB102 treatment (Experimental)
  Interventions: Drug: BB102

INTERVENTIONS:
Drug: BB102 — Oral BB102 Tablets in two dosage

SUMMARY:
This is a Phase 2 study to evaluate the efficacy and safety of BB102, a highly selective and potent FGFR4 inhibitor, as monotherapy in subjects with advanced or unresectable FGF19-overexpressing hepatocellular carcinoma. This study has two phase: dose escalation phase and expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18 years old, with no gender restrictions.
* (2) Disease progressed after receiving at least one anti-angiogenic and/or immune checkpoint inhibitor (including PD-1, PD-L1, CTLA-4) therapy, or the treatment is not tolerable.
* (3) Histologically confirmed primary HCC with FGF19 overexpression, which meets the Barcelona Clinic Liver Cancer (BCLC) staging criteria for patients with stage B suitable for systemic therapy or stage C.
* (4) At least one measurable lesion as defined by RECIST v1.1.
* (5) Eastern Cooperative Oncology Group (ECOG) score ≤1.
* (6) Expected survival ≥ 3 months.
* (7) Adequate organ function.
* (8) Female subjects of childbearing potential must have a negative pregnancy test prior to the first dose and are required to use effective contraception from signing the ICF until 6 months after the last dose of study treatment.
* (9) Fully informed of the study and voluntarily signed the informed consent form (ICF), and willing to follow and have the ability to complete all trial procedures.

Exclusion Criteria:

* (1) Use of systemic immunosuppressive or systemic cortisol (≥10 mg prednisone or other equivalent hormones) within 2 weeks.
* (2) Prior use of selective FGFR4 inhibitor therapy.
* (3) Use of Tyrosine kinase inhibitor within 2 weeks.
* (4) Use of systemic chemotherapy, radiotherapy (>30% bone marrow exposure), interventional embolization, ablation therapy and immunotherapycytotoxic chemotherapeutics within 4 weeks.
* (5) Use of other clinical investigational drug or therapy that was not marketed within 4 weeks.
* (6) The patient is receiving drugs or therapies prohibited in the protocol and cannot discontinue such use at least 7 days.
* (7) Pregnant or lactating females.
* (8) Presence of clinically significant gastrointestinal disorder that may affect the intake, transport, or absorption of the study drug at screening.
* (9) Patient with history of a second primary malignancy other than hepatocellular carcinoma within 5 years.
* (10) Presence of clinically symptomatic metastases to the central nervous system or meninges at screening, which, at the investigator's discretion, is not suitable for enrollment.
* (11) History of severe neurological or psychiatric disorders, including epilepsy, dementia, moderate to severe depression, etc.
* (12) Clinically significant and uncontrolled cardiovascular diseases.
* (13) Pulmonary embolism within 6 months.
* (14) Presence of uncontrollable infectious disease, congenital immunodeficiency disease,acquired immunodeficiency syndrome, syphilis, active hepatitis B, hepatitis C virus (HCV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From enrollment to the end of treatment assessed up to 12 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.

SECONDARY OUTCOMES:
Disease control rate (DCR) | From enrollment to the end of treatment assessed up to 12 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.
Duration of response (DOR) | From enrollment to the end of treatment assessed up to 12 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.
Progression-free survival (PFS) | From enrollment to the end of treatment assessed up to 12 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.
Time-To-Progression (TTP) | From enrollment to the end of treatment assessed up to 12 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.
Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | From enrollment to the end of treatment assessed up to 12 months
  AEs and SAEs will be characterized by type, seriousness, relationship to study treatment, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0) and timing.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Zhongshan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No